CLINICAL TRIAL: NCT04609579
Title: A Phase 1 Open-label Study of SNX281 Given as Monotherapy and in Combination With a Checkpoint Inhibitor in Subjects With Advanced Solid Tumors and Lymphoma
Brief Title: Study of SNX281 in Subjects With Advanced Solid Tumors and Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision (not due to safety concerns)
Sponsor: Stingthera, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SNX281-001; MK-3475-D44 (Other: Merck Sharp & Dohme LLC); KEYNOTE-D44 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2020-10-23; First posted 2020-10-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Advanced Solid Tumor; Advanced Lymphoma
Keywords: Stimulator of interferon genes; STING agonist; Ovarian Neoplasms; Colorectal Neoplasms; Microsatellite stable colorectal; Microsatellite instable colorectal; Lymphoma; B-Cell Lymphomas; Solid Tumor; Advanced Tumor
MeSH Terms: conditions — Bites and Stings; Ovarian Neoplasms; Colorectal Neoplasms; Lymphoma; Lymphoma, B-Cell | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SNX281 Monotherapy (Experimental): SNX281 will be administered weekly in Cycle 1 and then once every 3 weeks of each cycle thereafter for up to 6 cycles, or until disease progression or unacceptable toxicity occurs. Participants who are, in the opinion of the investigators, benefitting from treatment may be allowed to continue treatment with SNX281 beyond Cycle 6 with Sponsor approval. It is expected that up to approximately 66 participants will take part in this arm of the study.
  Subjects enrolled in the dose expansion phase of this arm may be eligible to add pembrolizumab (KEYTRUDA®) to their SNX281 therapy following identification of the maximum tolerated dose (MTD) or optimal dose of SNX281 in combination with pembrolizumab (KEYTRUDA®). Subjects must, in the opinion of the Investigator, have demonstrated tolerance to SNX281 and have experienced sub-optimal response to therapy (i.e., disease stability for 4 cycles or progression on treatment with SNX281 at any time).
  Interventions: Drug: SNX281
- SNX281 in Combination with pembrolizumab (KEYTRUDA®) (Experimental): SNX281 will be administered in 3 of the 4 weeks in Cycle 1 and then once every 3 weeks of each cycle thereafter. Participants will also receive pembrolizumab (KEYTRUDA®) once every cycle for up to 6 cycles. The combination of SNX281 and pembrolizumab (KEYTRUDA®) will be given for up to 6 cycles, or until disease progression or unacceptable toxicity occurs. Participants who are, in the opinion of the investigators, benefitting from treatment may be allowed to continue treatment with SNX281 and pembrolizumab (KEYTRUDA®) (or SNX281 alone) beyond Cycle 6 with Sponsor approval. It is expected that up to approximately 68 participants will take part in this arm of the study.
  Interventions: Drug: SNX281; Drug: pembrolizumab

INTERVENTIONS:
Drug: SNX281 — SNX281 will be administered as an intravenous infusion on Days 1, 8, and 15 in Cycle 1 and on Day 1 of each subsequent cycle thereafter of each 21-day cycle for up to 6 cycles, or until disease progression or unacceptable toxicity occurs. Cycle 1 length varies from 21 days in monotherapy arm to 28 days in the combination arm.
Drug: pembrolizumab — pembrolizumab (KEYTRUDA®) will be administered as an intravenous infusion on Day 8 in Cycle 1 (28-day cycle) and on Day 1 of each 21-day cycle thereafter for up to 6 cycles, or until disease progression or unacceptable toxicity occurs.
  Other Names: KEYTRUDA®
  Arms: SNX281 in Combination with pembrolizumab (KEYTRUDA®)

SUMMARY:
This clinical trial is evaluating a drug called SNX281 given by itself and in combination with pembrolizumab (KEYTRUDA®) in participants with advanced solid tumors and lymphoma. The main goals of this study are to:

* Find the recommended dose of SNX281 that can be given to participants safely alone and in combination with pembrolizumab (KEYTRUDA®).
* Learn more about the side effects and safety profile of SNX281 alone and in combination with pembrolizumab (KEYTRUDA®)
* Learn more about pharmacological characteristics of SNX281 alone and in combination with pembrolizumab (KEYTRUDA®)
* Learn more about effectiveness of SNX281 alone and in combination with pembrolizumab (KEYTRUDA®)

DETAILED DESCRIPTION:
SNX281 is a small molecule activator of the Stimulator of Interferon Genes (STING) protein, with good drug-like properties. Activation of STING initiates the innate immune response and enhances the adaptive immune response, which could potentially activate immune responses to tumors and enhance the response to certain immunotherapies.

This study is a phase I, first in human, open-label study of SNX281 conducted in subjects with advanced solid tumors and lymphomas. The study will comprise of two treatment arms: one evaluating SNX281 as a single-agent, and the other evaluating SNX281 in combination with pembrolizumab (KEYTRUDA®). Each treatment arm is designed to include a dose escalation phase followed by a dose expansion phase intended to establish the recommended Phase 2 dose (RP2D).

In the dose escalation phase of each treatment arm, successive cohorts of participants will receive increasing doses of SNX281 designed to determine the maximum tolerated dose (MTD), the dose with maximum pharmacologic activity, or the maximum feasible dose, as a single-agent and in combination with pembrolizumab (KEYTRUDA®).

The dose expansion phases of each treatment arm will begin following the determination of an MTD or alternative dose of SNX281 in each respective treatment arm. The single-agent treatment arm of SNX281 is planned to evaluate at least 2 expansion cohorts in ovarian cancer and colorectal carcinoma while the combination treatment arm of SNX281 and pembrolizumab (KEYTRUDA®) is planned to enroll subjects with advanced cancer who have relapsed on or have become refractory to prior immune checkpoint therapy given in an indicated setting.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet the following criteria in order to be included in the research study:

1. Written informed consent, according to local guidelines, signed and dated by the subject or by a legal guardian prior to the performance of any study-specific procedures, sampling, or analyses
2. At least 18 years-of-age at the time of signature of the informed consent form (ICF)
3. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1
4. Histological or cytological requirements as follows:

   a. Dose Escalation:

   i. All treatment arms: Subjects with histological or cytological documentation of advanced/recurrent solid tumors or lymphoma who have progressed on, are intolerant of, or are ineligible for existing standard therapies

   b. Dose Expansion:

   i. SNX281 Monotherapy: Subjects with histological or cytological documentation of advanced/recurrent ovarian or colorectal cancer who have progressed on, are intolerant of, or are ineligible for existing standard therapies. Subjects may be checkpoint inhibitor naïve. Subjects who qualify to add pembrolizumab (KEYTRUDA®) to their treatment regimen, must meet all medical eligibility requirements for receiving pembrolizumab (KEYTRUDA®) (see Inclusion Criteria 11).

   ii. SNX281 in Combination with pembrolizumab (KEYTRUDA®): Subjects with histological or cytological documentation of advanced/recurrent solid tumors or lymphoma who have relapsed on or are refractory to prior checkpoint inhibitor therapy given in an indicated setting. (Note: recruitment will be stopped in a given anatomical indication if no evidence of clinical response is observed in 15 subjects.)
5. Measurable or evaluable disease according to disease-specific tumor assessment criteria. Subjects in dose expansion portions of the study must have at least 1 measurable lesion that has not been previously irradiated, or has progressed after prior irradiation.
6. Subjects must have progressed on treatment with an anti-Programmed Cell Death Protein 1/Programmed Death-Ligand 1 (PD-1/L1) monoclonal antibody (mAb) administered either as monotherapy, or in combination with other checkpoint inhibitors or other therapies. PD-1/L1 treatment progression is defined by meeting all of the following criteria:

   1. Has received at least 2 doses of an approved anti-PD-1/L1 mAb.
   2. Has demonstrated disease progression (PD) after PD-1/L1 as defined by RECIST v1.1. The initial evidence of PD is to be confirmed by a second assessment no less than four weeks from the date of the first documented PD, in the absence of rapid clinical progression.
   3. Progressive disease has been documented within 12 weeks from the last dose of anti-PD-1/L1 mAb.

      * Progressive disease is determined according to iRECIST.
      * This determination is made by the Investigator. Once PD is confirmed, the initial date of PD documentation will be considered the date of disease progression.
7. Adequate organ function, defined as:

   a. Hematologic systems

   i. Absolute neutrophil count (ANC) ≥1.5 × 109/L

   ii. Hemoglobin ≥9 g/dL

   iii. Platelets ≥100 × 109/L

   b. Hepatic system

   i. Total bilirubin ≤1.5 × the upper limit of normal (ULN) (for subjects with Gilbert's Syndrome ≤3.0 × ULN [if direct bilirubin ≤35%])

   ii. Alanine aminotransferase and aspartate aminotransferase ≤2.5 × ULN; and for subjects with liver metastases ≤5.0 × ULN

   c. Renal system

   i. Estimated glomerular filtration rate (eGFR) by Cockcroft-Gault formula >50 mL/min

   d. Cardiac system

   i. Ejection fraction ≥50% by echocardiogram (ECHO) or multi-gated acquisition (MUGA) scan
8. A female subject is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP)
   2. A WOCBP who agrees to follow contraceptive guidance during the treatment period and for at least 6 months after the last dose of SNX281 and 120 days after the last dose of pembrolizumab (KEYTRUDA®), if applicable. WOCBP must have a negative urine pregnancy test within 72 hours prior to the first dose of study. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
9. Male subjects with female partners of childbearing potential are required to use two forms of acceptable contraception, including one barrier method, during their participation in the study and for 3 months following the last dose of SNX281, and for 120 days following the last dose of pembrolizumab (KEYTRUDA®). Male subjects must also refrain from donating sperm during their participation in the study and for 3 months following the last dose of SNX281 and 120 days after the last dose of pembrolizumab (KEYTRUDA®).
10. Life expectancy ≥12 weeks after the start of the treatment according to the Investigator's judgment.
11. Subjects considered for any combination of pembrolizumab (KEYTRUDA®) and SNX281 must meet, in the opinion of the Investigator, any additional criteria necessary for the safe and proper use of pembrolizumab (KEYTRUDA®).

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from study entry:

1. Malignancy other than the disease under study with the exception of those from which the subject has been disease-free for more than 2 years and not expected to affect the safety of the subject or the endpoints of the trial. Curatively treated non-melanoma skin cancer is permitted.
2. Symptomatic central nervous system (CNS) metastases or asymptomatic CNS metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during the study screening), clinically stable and without the requirement of steroid treatment for at least 14 days prior to first dose of study treatment. Subjects with carcinomatous meningitis or leptomeningeal spread are excluded regardless of clinical stability.
3. Active autoimmune disease that has required systemic disease modifying or immunosuppressive treatment within the last 2 years. Replacement therapy (e.g., thyroxine or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, insulin for type 1 diabetes, etc.) is permitted.
4. Concurrent medical conditions requiring the use of systemic immunosuppressive treatment within 28 days before the first dose of study treatment. Physiologic doses of corticosteroids (not exceeding 10 mg/day prednisone or equivalent) for treatment of endocrinopathies or steroids with minimal systemic absorption, including topical, inhaled, or intranasal corticosteroids may be continued if the subject is on a stable dose.
5. Current unstable liver or biliary disease per Investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis. Stable chronic liver disease (including Gilbert's syndrome or asymptomatic gallstones) or hepatobiliary involvement of malignancy is acceptable if subject otherwise meets entry criteria
6. History of vasculitis at any time prior to study treatment
7. Evidence or history of significant active bleeding or coagulation disorder that would compromise the subject's ability to adhere to the protocol.
8. Has a known history of HIV infection. No HIV testing is required unless mandated by local health authority(ies).
9. Has a known history of hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. No testing for hepatitis B or hepatitis C is required unless mandated by local health authority(ies).
10. Has an active infection requiring systemic therapy.
11. QT interval corrected for heart rate according to Fridericia's formula >480 msec by machine read or human over-read. Pre-existing bundle branch block is permitted at the Investigator's discretion.
12. Recent history (within the past 6 months) of acute diverticulitis, inflammatory bowel disease, intra-abdominal abscess, or gastrointestinal obstruction.
13. Recent history (within 4 weeks of starting study) of allergen desensitization therapy
14. History or evidence of cardiovascular risk including any of the following: recent (within the past 6 months) serious uncontrolled cardiac arrhythmia or clinically significant electrocardiogram (ECG) abnormalities including second degree (Type II) or third degree atrioventricular block; cardiomyopathy, myocardial infarction, acute coronary syndromes (including unstable angina pectoris), coronary angioplasty, stenting, or bypass grafting within the past 6 months before enrollment; congestive heart failure (Class II, III, or IV) as defined by the New York Heart Association functional classification system.
15. Recent (within the past 6 months) history of symptomatic pericarditis
16. History of idiopathic pulmonary fibrosis, interstitial lung disease, organizing pneumonia, non-infection pneumonitis that required steroids, or radiation pneumonitis. Note (SNX281 monotherapy only): post-radiation changes in the lung related to prior radiotherapy and/or asymptomatic radiation-induced pneumonitis not requiring treatment may be permitted if agreed upon by the Investigator and Sponsor
17. Symptomatic ascites or pleural effusions
18. Has known hypersensitivity (Grade ≥3) to pembrolizumab (KEYTRUDA®) and/or any of its excipients (for subjects receiving pembrolizumab (KEYTRUDA®) only).
19. Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with the subject's safety, obtaining informed consent, or compliance with study procedures
20. Prior treatment with the following agents:

    * Systemic stimulator of interferon genes (STING) agonist at any time (prior intra-tumoral STING agonist is acceptable)

      * Subjects treated in Treatment Arm 1 (SNX281 Monotherapy) who experience disease progression (PD) may be allowed to receive pembrolizumab (KEYTRUDA®) in combination with SNX281 with Sponsor approval
    * Anticancer therapy or investigational therapy within 28 days or 5 half-lives of the drug, whichever is shorter
    * PD-1, PD-L1, and cytotoxic T-lymphocyte-associated antigen 4 (CTLA-4) inhibitors within 28 days of the start of study treatment (SNX281 Monotherapy treatment arm only)
    * Received treatment with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX40, CD137), and was discontinued from that treatment due to Grade 3 or higher immune related AE for subjects receiving pembrolizumab (KEYTRUDA®) only.
    * Prior radiation therapy: permissible if at least 1 non-irradiated evaluable lesion is available for assessment according to disease-specific tumor response criteria, or if a solitary evaluable lesion was irradiated, objective progression of that lesion is documented. A washout period of at least 14 days before start of study treatment for radiation of any intended use to the extremities for bone metastases and 28 days for radiation to the chest or visceral organs is required. Participants must have recovered from all radiation-related toxicities, must not require corticosteroids, and must not have had radiation pneumonitis. For radiation to the brain, a washout period of at least 14 days for stereotactic body radiation therapy (SBRT) or stereotactic radiosurgery (SRS) and 28 days for whole brain radiotherapy (WBRT) is required. Palliative radiation with a 1-week washout is permissible at any other time for non-CNS disease before or during the study.
    * Subjects with mesothelioma, non-small cell lung cancer or small-cell lung cancer receiving pembrolizumab (KEYTRUDA®) with a history of radiation therapy to the lung >30Gy within 6 months of the first dose of pembrolizumab (KEYTRUDA®) are excluded.
    * Strong inhibitors and inducers of CYP3A4 must be discontinued 7 days or for a time equivalent to 5-half-lives of the medication (whichever is longer) prior to initiation of SNX281 treatment.
21. Receipt of any live vaccine within 30 days of the start of treatment
22. Prior allogeneic or autologous bone marrow transplantation or other solid organ transplantation
23. Toxicity from previous treatment including toxicity Grade ≥3 related to prior immunotherapy and that led to study treatment discontinuation; toxicity related to prior treatment that has not resolved to Grade ≤1 (except alopecia, hearing loss, or Grade ≤2 neuropathy or endocrinopathy managed with replacement therapy).
24. Received transfusion of blood products (including platelets or red blood cells) or administration of colony stimulating factors (including granulocyte colony stimulating factor, granulocyte-macrophage colony stimulating factor, and recombinant erythropoietin) within 7 days before the first dose of study treatment. Note: For subjects receiving pembrolizumab (KEYTRUDA®) only, packed red blood cell transfusions are not permitted within 2 weeks of treatment with pembrolizumab (KEYTRUDA®).
25. Major surgery ≤28 days before the first dose of study treatment. Subjects must have also fully recovered from any surgery (major or minor) and/or its complications before initiating treatment. Port-a-cath placement is permitted.
26. Active drug or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2024-01-06 (Actual); Study Completion 2024-01-06 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities to determine the maximum tolerated dose (MTD) and Recommended Phase 2 dose of SNX281 | Up to 28 Days
  Percentage of participants with dose limiting toxicities associated with SNX281 alone or SNX281 combined with pembrolizumab (KEYTRUDA®) during the first cycle. Toxicity will be assessed using the NCI CTCAE Version 5.0
Percentage of participants who experience adverse events and serious adverse events to determine safety and tolerability of SNX281 given as a single agent and in combination with pembrolizumab (KEYTRUDA®) | Up to 20 weeks
  Percentage of participants who experience adverse events and serious adverse events when given SNX281 as a single agent and in combination with pembrolizumab (KEYTRUDA®)

SECONDARY OUTCOMES:
Plasma concentration of SNX281 to characterize the pharmacokinetics (PK) parameters of SNX281 given as a single agent and in combination with pembrolizumab (KEYTRUDA®) | Up to 20 weeks
  Plasma concentration of SNX281 from all participants given as a single agent and in combination with pembrolizumab (KEYTRUDA®).
Plasma concentration of biomarker to determine pharmacodynamics (PD) response to SNX281 given as a single agent and in combination with pembrolizumab (KEYTRUDA®). | Up to 20 weeks
  Plasma concentration of biomarker from all participants receiving SNX281 as a single agent and in combination with pembrolizumab (KEYTRUDA®).
Objective response rate (ORR) to assess the clinical activity of SNX281 given as a single agent and in combination with pembrolizumab (KEYTRUDA®) | Up to 40 months
  Proportion of participants with confirmed complete response (CR) or partial response (PR) according to disease specific response criteria
  RECIST 1.1/iRECIST:
  A CR is the complete disappearance of all target and non-target lesions. A PR is a ≥30% decrease in the sum of diameters of target lesions from the baseline sum
  RECIL2017:
  A CR is the complete disappearance of all non-target/target lesions/all nodes with long axis <10 mm, or ≥30% decrease in the sum of longest diameters of target lesions (PR) with normalization of FDG-PET and no bone marrow involvement or appearance of new lesion. A PR is ≥30% decrease in the sum of longest diameters of target lesions, with positive FDG-PET with any bone marrow involvement and no appearance of new lesions and no progression of non-target lesions.
Duration of response (DoR) to assess the clinical activity of SNX281 given as a single agent and in combination with pembrolizumab (KEYTRUDA®) | Up to 40 months
  Defined as: Time from first documented response (CR or PR) to first evidence of progressive disease (PD) per RECIST 1.1 and RECIL 2017 or confirmed PD (iCPD) per iRECIST or death due to any cause.
  RECIST 1.1- PD: ≥20% increase in target lesions and ≥5mm from smallest sum, any new lesions, or unequivocal progression of non-target lesions.
  iRECIST- iCPD: Confirmation of further increase in tumor burden, compared to the last assessment where RECIST 1.1 definition of progression had been met, as evidenced by- ≥5 mm increase in progressed target lesion sum, increased size of previous unequivocally progressed non-target lesions, ≥5 mm increase in sum of previously identified new lesions, or new progression in target or non-target lesions or additional new lesions not previously identified.
  RECIL 2017- PD: New lesion appearance or ≥20% increase in sum of target lesions. If lymph N<15 mm post therapy,a ≥5 mm increase with longest diameter exceeds 15mm
Progression free survival (PFS) to assess the clinical activity of SNX281 given as a single agent and in combination with pembrolizumab (KEYTRUDA®) | Up to 40 months
  PFS: Time from the first day of study drug administration to disease progression (PD) as defined by disease-specific response criteria (RECIST 1.1, iRECIST, or RECIL2017), or death on study.
  RECIST 1.1- PD: ≥20% increase in target lesions sum and ≥5mm from smallest sum, any new lesions, or unequivocal progression of non-target lesions.
  iRECIST- iCPD: Confirmation of further increase in tumor burden, compared to the last assessment where RECIST 1.1 definition of progression had been met, as evidenced by- ≥5 mm increase in progressed target lesion sum, increased size of previous unequivocally progressed non-target lesions, ≥5 mm increase in sum of previously identified new lesions, or new progression in target or non-target lesions or additional new lesions not previously identified.
  RECIL 2017- PD: New lesion appearance or ≥20% increase in sum of longest diameters of target lesions. For lymph nodes measuring <15 mm post therapy, a ≥5 mm increase with longest diameter exceeds 15mm.
Overall survival (OS) to assess the clinical activity of SNX281 given as a single agent and in combination with pembrolizumab (KEYTRUDA®) | Up to 40 months
  Overall survival (OS) is defined as the time from the first day of study drug administration (Day 1) to death
Disease control rate (DCR) to assess the clinical activity of SNX281 given as a single agent and in combination with pembrolizumab (KEYTRUDA®) | Up to 40 months
  DCR is: Proportion of subjects who achieved either a complete response (CR), partial response (PR), or stable disease (SD) at their first scheduled disease assessment according to disease-specific response criteria.
  RECIST 1.1/iRECIST CR: disappearance of all target/non-target lesions. PR: ≥30% decrease in the sum of diameters of target lesions from baseline sum. SD: Neither sufficient shrinkage to qualify for a PR nor sufficient increase in lesions for a PD
  RECIL2017 CR: Disappearance of all target/nodal lesions or ≥30% decrease in the sum of longest diameters of target lesions with normal FDG-PET and no bone marrow (BM) involvement or new lesion.
  PR: ≥30% decrease in the sum of longest diameters of target lesions with positive FDG-PET with any BM involvement and no new lesion.
  SD: Less than 10% decrease or up to 20% increase in the sum of longest diameter of target lesions with any FDG-PET result or any bone marrow involvement and no appearance of new lesion

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Johnson, MD, Study Chair — SCRI Development Innovations, LLC
Locations (4):
- United States (4):
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Florida Cancer Specialists, Sarasota, Florida
  - Thomas Jefferson University, Sidney Kimmel Cancer Center, Philadelphia, Pennsylvania
  - Tennessee Oncology, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No